CLINICAL TRIAL: NCT02571439
Title: A Randomized Controlled Trial of Surgical TAP-block After Cesarean Delivery: a Cost-effective Alternative to the Conventional TAP-block
Brief Title: Comparative Study of Two Different Techniques to Perform TAP-blocks
Acronym: Surgical-TAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, kalpana tyagaraj, MD, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 2014-08-05
Record Dates: First submitted 2014-08-16; First posted 2015-10-08 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: POSTOPERATIVE PAIN
Keywords: TAP block, post-cesarean analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical TAP block (Experimental): surgeon administered intraoperative TAP block using 0.5% ropivacaine
  Interventions: Procedure: Surgical TAP block; Drug: 0.5% ropivacaine
- Conventional TAP block (Active Comparator): Conventional, Anesthesiologist administered post-operative TAP block using 0.5% ropivacaine
  Interventions: Procedure: Conventional TAP block; Drug: 0.5% ropivacaine

INTERVENTIONS:
Procedure: Surgical TAP block — surgeon administered TAP block
  Arms: Surgical TAP block
Procedure: Conventional TAP block — Anesthesiologist administered TAP block
  Arms: Conventional TAP block
Drug: 0.5% ropivacaine — 20ml of 0.5% ropivacaine is used to perform the TAP block
  Other Names: Naropin

SUMMARY:
The TAP is a space between the muscle layers of the abdominal wall that houses nerves supplying the abdominal skin. Injecting the local anesthetic ropivacaine into this space will block these nerves and prevent pain following c-section. The investigators will compare two different approaches to injecting the local anesthetic in this space. Conventionally, the block is done after surgery is completed and the abdomen is closed. The anesthesiologist introduces a needle through the abdominal wall skin under ultrasound guidance to reach the TAP space and the drug is injected. Since the TAP layer is one of the deeper layers of the abdominal (belly) wall and is closer to the inside of the abdomen than to the outside (skin), injecting from the inner aspect of the abdominal wall during the surgery is easier and quicker to perform than the conventional block and does not require ultrasound guidance as there is no risk of injury to abdominal organs like the liver.

With this research the investigators attempt to prove that surgically administered TAP blocks take 25% less time to perform compared to the conventionally administered TAP block for post cesarean section pain relief. Surgical TAP blocks are also more cost-effective as in addition to reduced OR time, they are safer and do not require skilled operator and specialized equipment. Secondary outcomes will include total time spent in the Operating room, presence and severity of postoperative pain, time to first request for pain medication, total postoperative narcotic consumption in 48 hours after surgery and side effects.

DETAILED DESCRIPTION:
The investigators propose to perform a prospective randomized trial of the surgically administered TAP block as compared to the conventional TAP block. The investigators will recruit women undergoing scheduled cesarean delivery under neuraxial anesthesia. Participants will be recruited in the labor and delivery of Maimonides Medical Center. Written informed consent will be obtained from the patients in a standardized consent form which explains the voluntary nature of the study, benefits and risks of both procedures and alternatives.

Sample size calculation: Estimates of time taken to perform the anesthetic block in our set up was an average of 10 minutes and standard deviation of 3.75 minutes (range 5-20min). The number of participants necessary to detect a 25% reduction in the time taken to perform the block with a power of 80% and α=0.05 was 36 patients in each group and a total of 72 patients. Allowing for a 15% dropout rate will require 42 patients to be recruited in each group and a total of 84 patients. The investigators will initially conduct a pilot study with the first five patients. Patients will undergo stratified block randomization to control for BMI (BMI<40 and BMI> or =40), complexity of surgery based on number of previous uterine scars (< or = 2previous scars, 3 or more previous scars) Anesthetic regimen: Cesarean sections will be performed under neuraxial anesthesia- spinal, epidural and combined spinal-epidural. Standard dosing of local anesthetic will be used in all patients. Patients receiving supplemental short acting non-opioid medication (eg: ketamine) intraoperatively will be included but patients converted to general anesthesia will be excluded.

TAP Block: The conventional TAP block is performed after the skin is closed at the completion of surgery and after the dressing is applied. The abdomen will be prepped and draped in a sterile fashion and the block performed under sonographic guidance at the level of the umbilicus in the anterior axillary line. A blunt tip 21G needle will be used to perform the block and 20ml of 0.5% ropivacaine will be injected after confirming the location of the needle on sonogram. Similar procedure will be repeated on the other side. The surgical TAP block will be performed by a technique adapted from the description by DJ Owen et al (Owen DJ, 2011). After uterine closure is completed and good hemostasis has been secured, the abdominal wall on the side away from the surgeon will be retracted superiorly by the surgical assistant and the surgeon will palpate the lateral border of the rectus muscle. The block will be performed lateral to the rectus muscle in order to avoid injury to the inferior epigastric vessels. Safe access to the TAP plane will be achieved by inserting a blunt needle through the parietal peritoneum and transverse abdominis muscle during which time there is an appreciable loss of resistance ('one pop'). The needle and local anesthetic drug used is identical to that of the conventional TAP block. After careful aspiration, to ensure no vascular injury has occurred, 1 ml of the anesthetic solution is introduced slowly. The presence of substantial resistance to injection or a bleb formation (at the peritoneal site) suggests incorrect needle tip position, resulting in needle repositioning by advancement or retraction as required. The surgeon will feel the expanse of this plane after a significant volume is injected with very little resistance. The surgical TAP block will then be performed on the other side in a similar manner except the surgeon will switch sides with the assistant for better visualization while performing the block. Following the block, the rectus sheath and skin will be closed in the usual manner.

Blinding: The patient and the operator assessing postoperative outcomes measures (pain, analgesic requirements, side effects and patient satisfaction) will be blinded to the allocation. The investigator assessing primary outcome (time taken to perform the block) cannot be blinded due to the nature of the study but will be an independent observer and not the surgeon or anesthesiologist performing the procedures. The investigators will have two independent observers collecting data on time outcomes to reduce error and also have the procedure filmed on a random sample of 10% of patients to verify the times assigned by the study personnel.

Postoperative: Each woman will be prescribed a standard analgesic regimen of toradol 30mg IV every 8 hours and IV Tylenol 1000mg every 6 hours as needed. Morphine PCA will also be available for pain not controlled with toradol and Tylenol. The presence and severity of postoperative pain, sedation, nausea/vomiting, and respiratory depression will be assessed postoperatively at 4, 8, 24 and 48 hours by an investigator blinded to group allocation. The time to first request for rescue analgesia and total consumption of opioid and non-opioid pain medication in 48 hours will also be recorded. The severity of pain at rest and on coughing will be as assessed using a 10-cm visual analog scale (0 no pain and 10 worst imaginable pain). Presence of side effects like nausea/vomiting, sedation and itching will be recorded.

Outcomes: The primary outcome is the time taken to perform the block (conventional TAP block and the surgical TAP block). Secondary outcomes include time components (total time spent in the Operating room, time from uterine closure with hemostasis to exit from OR) and postoperative outcomes (presence and severity of postoperative pain, time to first request for rescue analgesic, total consumption of pain medication 48 hours after surgery, sedation, postoperative nausea/vomiting, itching).

Statistical analysis: Standard descriptive statistics will be used and mean or median will be used to describe data depending on whether the assumptions of normality are violated. For the primary outcome which is time taken to perform the block, student t test or other appropriate nonparametric test to compare differences between the two groups will be performed. An intention to treat analysis will be performed. All calculations will be done using SPSS software. Senior biostatistician Dr Peter Homel will be performing the analysis.

The study will be suspended on Fridays, Saturdays, Sundays, and observed religious holidays. Physicians and nursing staff from the Department of Anesthesiology and Obstetrics blinded to the dose of ropivacaine administered will collect data at 4, 8, 24, and 48 hours after cesarean section through verbal interaction of the staff with the patients. The patients' answers will be recorded on data collection sheets and placed in the chart for future analysis by the principal and co-investigators, and other physicians and nursing staff affiliated with the Departments of Anesthesiology and Obstetrics. For quality control there will be a bimonthly review of data collected to ensure the integrity and completeness of the information collected.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit women undergoing scheduled cesarean delivery under neuraxial anesthesia

Exclusion Criteria:

* Age less than 18 years
* We will limit recruitment to women able to speak atleast one of the following languages: English, Spanish, Chinese, Russian
* Chronic pain syndrome
* Opioid dependence
* Allergy to local anesthetic
* Vertical skin incision
* Sepsis at the site of injection
* Converted to general anesthesia
* Any complicated procedures including blood loss more than 2000ml and duration of surgery more than 2 hours.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Tyagaraj, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to recruitment proceeding slower than expected and study personnel relocating from the study site, we closed the study before recruitment of planned number of subjects
Period: Overall Study
Arm/Group | Surgical TAP Block | Conventional TAP Block
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Surgical TAP: Intra-operative TAP block
- Conventional TAP: Percutaneous ultrasound guided TAP block
- Total: Total of all reporting groups
Arm/Group | Surgical TAP | Conventional TAP | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (4.0) | 32.2 (5.4) | 30.7 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 21 | 41
BMI [Mean (Standard Deviation); unit: Kg/m^2] — Kg/m2
  Kg/m^2 | 31.2 (5.6) | 30.7 (6.5) | 31.0 (6.0)
Previous abdominal surgery [Count of Participants; unit: Participants]
  Yes | 17 | 16 | 33
  No | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Time Taken to Perform the Block
Description: Two independent observers (who are not the surgeon or anesthesiologist performing the procedures) will collect data on time outcomes to reduce error and the procedure will be filmed on a random sample of 10% of patients to verify the times assigned by the study personnel. Filming will be started after the patient is draped so that the patients face is not in the recording.
Time Frame: The time taken to perform the block in the operating room is measured, upto 60 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
minutes | 2.4 (0.5) | 12.1 (5.1)
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Time From Delivery of Neonate to Ready to Exit Operating Room
Description: as for outcome 1
Time Frame: Time measures will be recorded in the operating room, upto 6 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
minutes | 55.3 (10.2) | 77.9 (18.9)
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Severity of Postoperative Pain at Rest
Description: postoperative pain will be assessed using the visual analog scale postoperatively at 4 hours after surgery. visual analog pain scale is a response scale to measure pain with a score of 0 representing no pain and a score of 10 representing the worst pain imaginable. The minimum value was 0 for no pain and maximum value was 10 for the worst pain imaginable. The responses are whole numbers ranging from 0 to 10 with increasing numbers representing increasing pain.
Time Frame: 4 hours after surgery
Measure: Median (Inter-Quartile Range); unit: Numerical rating scale for pain
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
Numerical rating scale for pain | 4 [2 to 5] | 3 [2 to 6]
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p = 0.61, Kruskal-Wallis

4. Secondary Outcome: Severity of Postoperative Pain at Rest
Description: postoperative pain will be assessed using the visual analog scale postoperatively at 8 hours after surgery. v
Time Frame: 8 hours after surgery
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
Units on a scale | 4 [2 to 5] | 3 [2 to 5]
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p = 0.46, Kruskal-Wallis

5. Secondary Outcome: Severity of Postoperative Pain at Rest
Description: postoperative pain will be assessed using the visual analog scale postoperatively at 24 hours after surgery. v
Time Frame: 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
Units on a scale | 2 [0 to 4] | 3 [1 to 4]
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p = 0.33, Kruskal-Wallis

6. Secondary Outcome: Severity of Postoperative Pain at Rest
Description: postoperative pain will be assessed using the visual analog scale postoperatively at 48 hours after surgery.
Time Frame: 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
Units on a scale | 2 [0 to 5] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p = 0.13, Kruskal-Wallis

7. Other Pre Specified Outcome: Total Narcotic Consumption
Description: Total narcotic consumption, measured in mg of morphine 24 hours after surgery
Time Frame: 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mg of morphine
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
mg of morphine | 28 [20 to 51] | 25 [9 to 38]
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p = 0.17, Kruskal-Wallis

8. Other Pre Specified Outcome: Sedation
Description: sedation will be assessed postoperatively on a scale of 0 to 10. The minimum value was 0 for not sedated or awake and maximum value was 10 for extremely sedated. The responses are whole numbers ranging from 0 to 10 with increasing numbers representing increasing sedation.
Time Frame: up to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: scale of 0-10
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
scale of 0-10 | 2.5 [0 to 7.5] | 3 [0 to 6]
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p = 0.87, Kruskal-Wallis

9. Other Pre Specified Outcome: Number of Participants With Postoperative Nausea/Vomiting
Description: outcomes will be assessed postoperatively as number of patients with postoperative nausea/vomiting "present" or "not present" at 24 hours after surgery
Time Frame: up to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
Participants | 3 | 1
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p = 0.27, Chi-squared

10. Other Pre Specified Outcome: Itching.
Description: Itching will be assessed postoperatively on a scale of 0 to 10 at 24 hours after surgery. The minimum value was 0 for no itching and maximum value was 10 for severe itching. The responses are whole numbers ranging from 0 to 10 with increasing numbers representing increasing itching.
Time Frame: up to 24 hours after surgery
Measure: Median (Inter-Quartile Range); unit: scale of 0-10
Arm/Group | Surgical TAP Block | Conventional TAP Block
Number analyzed (Participants) | 20 | 21
scale of 0-10 | 0 [0 to 2.5] | 0 [0 to 3]
Statistical Analysis 1: Comparison: Surgical TAP Block vs Conventional TAP Block; Test type: Other; p = 0.91, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | Surgical TAP Block | Conventional TAP Block
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

LIMITATIONS AND CAVEATS:
Personnel in OR could not be blinded due to nature of study. Personnel providing postop care and collecting postop data were blinded. Our study was not powered to explore the secondary outcomes; a larger study is needed to confirm those findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No